CLINICAL TRIAL: NCT00700882
Title: A Phase II Trial of Dasatinib in KIT-Positive Patients With Unresectable Locally Advanced or Stage IV Mucosal, Acral and Vulvovaginal Melanomas
Brief Title: Dasatinib in Treating Patients With Locally Advanced or Metastatic Mucosal Melanoma, Acral Melanoma, or Vulvovaginal Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2607; E2607 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; acral melanoma; mucosal melanoma; vulvovaginal melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dasatinib (Experimental): Patients receive oral dasatinib at 70 mg twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Patients receive oral dasatinib at 70 mg twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Other Names: Sprycel; BMS-354825

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well dasatinib works in treating patients with locally advanced or metastatic mucosal melanoma or acral melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the objective tumor response rate in patients with KIT-positive, unresectable, locally advanced or metastatic acral or mucosal melanoma treated with dasatinib monotherapy.

Secondary

* To estimate the response duration in patients treated with this drug.
* To estimate the progression-free survival of patients treated with this drug.
* To evaluate the safety profile of this drug in these patients.
* To evaluate the PDGFR expression and activation of Src family kinases in tumor samples and correlate these parameters with response to treatment.

OUTLINE: This is a multicenter study.

Patients receive oral dasatinib twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Tissue samples may be collected from some patients for correlative studies.

After completion of study therapy, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria for Pre-Registration (Step 0):

* Histologically or cytologically confirmed melanoma of 1 of the following subtypes:

  * Acral melanoma (defined as occurring on the palms, soles, or subungual sites)
  * Melanoma arising from the vagina and/or vulva
  * Melanoma arising on other mucosal surface (not vagina or vulva)
* Unresectable locally advanced or metastatic disease
* c-KIT mutation identified by polymerase chain reaction (PCR) and sequencing meeting 1 of the following criteria:

  * At least 1 mutation in exon 9, 11, 13, 17, or 18
  * At least 1 mutation in an exon not listed above and approved by central reviewer
* Metastatic tumor blocks are required for the evaluation of KIT mutations or amplifications
* Prior radiotherapy to a measurable lesion allowed provided there is radiographic evidence of progression of that lesion
* No other concurrent malignancies except basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, ductal or lobular carcinoma in situ of the breast, or other malignancies from which the patient has been continuously disease-free for ≥ 5 years
* ECOG performance status 0-1

Exclusion Criteria for Pre-Registration (Step 0):

* Prior treatment with targeted therapies directed to c-KIT/PDGFR (e.g., imatinib or sunitinib)
* Ocular melanoma
* Evidence of bleeding diathesis
* Clinically significant psychiatric illness or social situations that would limit compliance with study requirements
* Clinically significant cardiovascular disease including the following:

  * Myocardial infarction or ventricular tachyarrhythmia within 6 months
  * Prolonged QTc >480 msec (Fridericia correction)
  * Ejection fraction less than institutional normal
  * Major conduction abnormality (unless a cardiac pacemaker is present)
  * Patients with any cardiopulmonary symptoms of unknown cause (e.g., shortness of breath, chest pain, etc.) are to be evaluated by a baseline echocardiogram with or without stress test as needed in addition to electrocardiogram (EKG) to rule out QTc prolongation
  * Patients with underlying cardiopulmonary dysfunction are excluded from the study

Inclusion Criteria for Registration (Step 1):

* Meeting the eligibility criteria for pre-registration (Step 0)
* The melanoma must harbor a c-KIT mutation determined by PCR and sequencing as defined in the protocol either by local assessment or Massachusetts General Hospital (MGH)
* Measurable disease, defined as at least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* At least 4 weeks since prior chemotherapy, radiotherapy or immunotherapy and the beginning of protocol therapy and the patient must have recovered from toxicity due to the previous therapy
* History or clinical evidence of brain metastasis allowed provided the following criteria are met:

  * Completed radiotherapy or surgical treatment of brain lesions and there is no evidence of central nervous system (CNS) progression for ≥ 8 weeks
  * Must not require corticosteroids for treatment of cerebral edema from brain metastases
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients must have the following within 4 weeks of registration:

  * computed tomography (CT) chest with intravenous (IV) and oral agent
  * CT pelvis/abdomen with IV and oral agent
  * MRI brain with gadolinium
* Baseline bone scan required for patients with known bone metastases, elevated alkaline phosphatase, or symptoms raising suspicion of bone metastases
* White blood count (WBC) ≥ 3,000/mm³
* Absolute granulocyte count (AGC) ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 times upper limit of normal (ULN) OR creatinine clearance (CrCl) ≥ 40 mL/min
* Total bilirubin ≤ 1.5 times ULN (< 3.0 times ULN in the presence of Gilbert disease)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN (≤ 5.0 times ULN in the presence of liver metastases)
* Serum potassium and magnesium normal (repletion allowed)
* Total serum calcium or ionized calcium ≥ institutional lower limit of normal
* International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) wtihin normal limits

  * Therapeutic anticoagulation with warfarin allowed provided INR ≤ 1.5 or PTT normal prior to initiating anticoagulation therapy

Exclusion Criteria for Registration (Step 1):

* Pregnant or nursing
* Concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (i.e., phenytoin, carbamazepine, or phenobarbital), rifampin, or Hypericum perforatum (St. John wort)
* Uncontrolled hypertension, defined as systolic blood pressure ≥ 150 mm Hg or diastolic blood pressure ≥ 90 mm Hg

  * Hypertension that is adequately controlled with medication allowed
* QTc prolongation, defined as a QTc interval ≥ 450 msecs
* Serious intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-07-02 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald P. Lawrence, MD, Study Chair — Massachusetts General Hospital; Kevin Kalinsky, MD, Principal Investigator — Tufts Medical Center Cancer Center
Locations (153):
- United States (153):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford Cancer Center, Stanford, California
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Parvin Radiation Oncology, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Kalinsky K, Lee S, Rubin KM, Lawrence DP, Iafrarte AJ, Borger DR, Margolin KA, Leitao MM Jr, Tarhini AA, Koon HB, Pecora AL, Jaslowski AJ, Cohen GI, Kuzel TM, Lao CD, Kirkwood JM. A phase 2 trial of dasatinib in patients with locally advanced or stage IV mucosal, acral, or vulvovaginal melanoma: A trial of the ECOG-ACRIN Cancer Research Group (E2607). Cancer. 2017 Jul 15;123(14):2688-2697. doi: 10.1002/cncr.30663. Epub 2017 Mar 23. PMID 28334439
- [Derived] Kalinsky K, Hong F, McCourt CK, Sachdev JC, Mitchell EP, Zwiebel JA, Doyle LA, McShane LM, Li S, Gray RJ, Rubinstein LV, Patton D, Williams PM, Hamilton SR, Conley BA, O'Dwyer PJ, Harris LN, Arteaga CL, Chen AP, Flaherty KT. Effect of Capivasertib in Patients With an AKT1 E17K-Mutated Tumor: NCI-MATCH Subprotocol EAY131-Y Nonrandomized Trial. JAMA Oncol. 2021 Feb 1;7(2):271-278. doi: 10.1001/jamaoncol.2020.6741. PMID 33377972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 81 patients were accrued between May 1, 2009 and December 28, 2015 and the study was closed due to slow accrual. The first patient was accrued on July 2, 2009.
Period: Overall Study
Arm/Group | Dasatinib
Started | 81
Received Protocol Therapy | 75
Eligible and Treated Patients | 73
Eligible, Treated and KIT+ Patients | 22
Eligible and Treated Patients With Objective Response | 7
Completed | 22
Not Completed | 59
Not completed — Never received treatment | 6
Not completed — Ineligible | 2
Not completed — No KIT mutation | 51

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Dasatinib
Number analyzed (Participants) | 73
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 66
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Among KIT-positive Patients
Description: Objective response is defined as complete response (CR) or partial response (PR) per Solid Tumor Response Criteria (RECIST). Complete response is defined as disappearance of all target and non-target lesions. Partial response is defined as at least 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Every 6 weeks; up to 5 years
Population: eligible and treated KIT-positive patients
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 22
proportion of participants | 0.182 [0.104 to 0.466]

2. Secondary Outcome: Duration of Response for Dasatinib Monotherapy in This Patient Population
Description: Duration of response is defined as the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the first date that progressive disease is objectively documented, taking as reference the smallest measurements recorded since treatment started. Progressive disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Time Frame: Every 6 weeks; up to 5 years
Population: Only eligible and treated patients with objective response (complete response or partial response) are included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 7
months | 4.2 [0 to 17.1]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to development of progressive disease. Patients without documented progressive disease are censored at the date of last disease assessment. Progressive disease is defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s).
Time Frame: Every 6 weeks; up to 5 years
Population: Only eligible and treated patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dasatinib
Number analyzed (Participants) | 73
months | 2.1 [1.5 to 2.9]

4. Other Pre Specified Outcome: To Evaluate the PDGFR Expression, and Activation of Src Family Kinases in Tumor Samples and Correlate These Parameters With Response to Treatment.
Description: as for outcome 1
Time Frame: Every 6 weeks; up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Description: Adverse events were evaluated among all treated patients, regardless of eligibility.
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 15/75
Serious Adverse Events (participants affected / at risk) | 35/75
Other Adverse Events (participants affected / at risk) | 54/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=75)
Anemia (Blood and lymphatic system disorders) | 5
Chest pain - cardiac (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 10
Diarrhea (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Cardiac troponin I increased (Investigations) | 1
Cardiac troponin T increased (Investigations) | 1
INR increased (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=75)
Anemia (Blood and lymphatic system disorders) | 24
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 24
Diarrhea (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 6
Aspartate aminotransferase increased (Investigations) | 8
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less